CLINICAL TRIAL: NCT04073212
Title: Dry Needling and Heavy Slow Load Exercise Versus Traditional Physical Therapy in the Treatment of Individuals With Bicipital Tendinopathy; A Pilot Study
Brief Title: Dry Needling and Exercise Versus Traditional Physical Therapy for Biceps Tendinitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to inability to recruit and enroll during COVID-19
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Newcastle, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-2791
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Bicep Tendinitis; Biceps; Tenosynovitis; Bicipital Tendinitis, Left Shoulder; Bicipital Tendinitis, Right Shoulder; Bicipital Tendinitis, Unspecified Shoulder; Biceps Tendon Disorder
Keywords: dry needling; eccentric exercise; concentric exercise; physical therapy; heavy slow load exercise
MeSH Terms: conditions — Tenosynovitis | interventions — Dry Needling; Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 arms or treatment groups
Who Masked: Outcomes Assessor
Masking Description: Concealed allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention 1 DN+HSLE (Experimental): Patients in the intervention 1 Dry Needling (DN)+heavy Slow Load Exercise (HSLE) group will attend physical therapy one to two sessions per week for up to 4 weeks for a total of 6 sessions. Each treatment session will last for a total of 45 minutes. A standardized physical therapy program will be used and will include soft tissue mobilization to the shoulder and biceps tendon followed by DN, HSLE and a standardized shoulder strengthening exercise program.
  Interventions: Other: Dry Needling; Other: Heavy Slow Load Exercise; Other: Rotator cuff and scapular stabilization exercise program; Other: Soft tissue mobilization
- Intervention 2 Control (Active Comparator): Patients in the control group will attend physical therapy one to two sessions per week for up to 4 weeks for a total of 6 sessions. Each treatment session will last for a total of 45 minutes. A standardized physical therapy program will be used and will include soft tissue mobilization to the shoulder and biceps tendon and a standardized exercise program. Dry needling nor heavy slow load exercise will not be integrated into the "control" plan of care.
  Interventions: Other: Rotator cuff and scapular stabilization exercise program; Other: Soft tissue mobilization

INTERVENTIONS:
Other: Dry Needling — Dry needling directly to the long head of the biceps tendon. The DN will be performed with disposable stainless-steel needles (.3 X 40mm; Seirin; Weymouth, MA) inserted into the skin over the most painful and/or thickened areas of the tendon, confirmed with palpation. Prior to insertion of the needle the overlying skin will be cleaned with alcohol. The needle will be inserted into the tendon. The technique will be a fast-in and fast-out technique described by Chiavaras et al.26 for 20-30 repetitions per session in up to 3 areas. An eccentric-concentric exercise program of the biceps muscle/tendon will follow each DN session and will be performed daily for the course of treatment and will be performed as described by McDevitt et al.
  Other Names: Manual Therapy
  Arms: Intervention 1 DN+HSLE
Other: Heavy Slow Load Exercise — Eccentric exercise protocols have been found to be an effective treatment for tendinopathies of the upper and lower extremities and recent evidence supports heavy slow resistance training (including the addition of a concentric phase) as having better outcomes over eccentric exercise alone. Patients will use 1-5 pound weights to perform slow and controlled concentric and eccentric exercise to biceps muscle.
  Other Names: Therapeutic Exercise
  Arms: Intervention 1 DN+HSLE
Other: Rotator cuff and scapular stabilization exercise program — Both groups will be treated with a stretching and strengthening program. The rotator cuff and scapular stabilization strengthening and flexibility program used in this study has 3 phases and patients progress in phases based on their ability to perform a number of exercises using theraband or body weight resistance.
  Other Names: Therapeutic Exercise
Other: Soft tissue mobilization — Both groups will receive soft tissue mobilization to the anterior shoulder.
  Other Names: Manual Therapy

SUMMARY:
The aim of the research is to determine if participants who receive physical therapy (physiotherapy) including soft tissue mobilization, dry needling, Heavy slow load (eccentric-concentric) exercise (with hand weights specific to the biceps muscle) and a comprehensive rotator cuff and scapular stabilization program achieve greater reductions in pain and disability in the short (3-4 weeks) and long term (6 months) compared to those who receive soft tissue mobilization and a comprehensive rotator cuff and scapular stabilization program. Both treatment approaches are within the standard of care for physical therapists, the aim being to determine the most effective treatment approach. Study participants will be recruited form clinicians and flyers within the university/hospital organization where the study is taking place. Participants will be asked to attend 6 physical therapy visits and complete 6 surveys about their pain and disability.

DETAILED DESCRIPTION:
The overall purpose of the pilot study is to test the feasibility of methods and procedures for later use to conduct a large study to determine if patients who receive physical therapy including dry needling, heavy slow load exercise and a comprehensive rotator cuff and scapular stabilization program achieve greater reductions in pain and disability in the short (4 weeks) and long term (6 months) compared to those who receive soft tissue mobilization and a comprehensive rotator cuff and scapular stabilization program. A secondary purpose is to search for possible effects and associations between variables that may be worth following up in a subsequent, larger study.

Hypothesis: 1) Individuals with biceps tendinopathy who receive an intervention of soft tissue mobilization, dry needling (DN), heavy slow load exercise (HSLE) and a comprehensive rotator cuff and scapular stabilization program will demonstrate significant differences in disability and pain scores compared to the control group as measured by the:

1. American Shoulder and Elbow Surgeons Standardized Shoulder Form (ASES.) This improvement will be a minimum mean difference of 8 points (standard deviation, 12 points) between groups which would indicate a clinically meaningful improvement.
2. Disabilities of the Arm Shoulder and Hand (DASH)
3. Patient Specific Functional Scale (PSFS)
4. Numeric Pain Rating Score (NPRS)
5. Shoulder Hand and Disability Index (SPADI)

Inclusion Criteria:

1. Age 18-64 years old
2. Primary complaint of anterior shoulder pain in the area of the LHBT
3. Clinical exam findings (must have positive findings for at least 1/2 of the following). Several tests have been described for isolating pathology of the LHBT, however literature has shown that none of these tests are specific enough in isolation to confirm the diagnosis9 and Speed's test and Yergason's test do not perform consistently and they do not generate a large change in post-test probability.59 Additionally, better diagnostic utility is accomplished when 2 highly sensitive tests and one highly specific test60 however, Speed's and Yergason's tests are both specific. Therefore, it was decided that 1/2 specific tests would still be potentially inclusive of the pathology since neither of the tests is specific enough to confirm diagnosis either combined or in isolation.9,61 A test cluster of Speed's test combined with biceps palpation was reported to have a sensitivity of 68% and a specificity of 49%.12

   a. Speed's i. Speed's test (sensitivity 32%, specificity 75% for biceps pathology) was performed by having the clinician extend the elbow, supinate the arm and elevate the humerus with resistance to approximately 60 degrees; a positive test is pain in the bicipital groove region.62-64 b. Yergason's i. Yergason's test (sensitivity 43%, specificity 79% for biceps pathology) was performed by having the clinician flex the elbow to 90 degrees with a pronated forearm. The clinician would then have the patient resist supination with pressure at the patient's wrist. A positive test is pain in the area of the bicipital groove.65,66
4. Pain with palpation in area of the LHBT. Positive pain with palpation in the region of the LHBT and intertubercular groove has been found to be diagnostic for bicipital tendinopathy (sensitivity 27-53%, specificity 54-66%). 9,41,67
5. Patient identification of pain in the area of the proximal biceps tendon.8,9
6. NPRS of at least 3/10 at worst in the past week a. A minimal score of 3/10 was utilized in a case series on individuals with bicipital tendinopathy who were treated with DN and eccentric-concentric exercise.30 In addition, anecdotally these patients tend to have low but persistent pain.

Exclusion Criteria:

1. History of biceps tendon injection in the past 3 months
2. History of rotator cuff surgery
3. History of biceps tenodesis or tenotomy
4. History of bleeding disorder or anti-coagulation therapy
5. Diagnosis of adhesive capsulitis (as defined by 50% loss of range of motion in 2 out of 3 of the following motions: Shoulder flexion, abduction and external rotation)
6. Known underlying non-modifiable medical condition (e.g. tumor, fracture, metabolic disease)
7. Two or more positive neurological signs consistent with nerve root compression
8. Known allergy to metal
9. Participant reported aversion to needles

Participants will be randomized to 1 of 2 groups;

1. Dry Needling/Heavy Slow Load Exercise
2. Heavy Slow Load Exercise (Control)

Patients in the intervention 1 (DN+HSLE) group will attend physical therapy one to two sessions per week for up to 4 weeks for a total of 6 sessions. Each treatment session will last for a total of 45 minutes. A standardized physical therapy program will be used and will include soft tissue mobilization to the shoulder and biceps tendon followed by DN, HSLE and a standardized exercise program. The DN will be performed with disposable stainless-steel needles (.3 X 40mm; Seirin; Weymouth, MA) inserted into the skin over the most painful and/or thickened areas of the tendon, confirmed with palpation. Prior to insertion of the needle the overlying skin will be cleaned with alcohol. The needle will be inserted into the tendon. The technique will be a fast-in and fast-out technique described by Chiavaras et al.26 for 20-30 repetitions per session in up to 3 areas. A HSLE program of the biceps muscle/tendon will follow each DN session and will be performed daily for the course of treatment and will be performed as described by McDevitt et al.30

Participants in the control group will attend physical therapy one to two sessions per week for up to 4 weeks for a total of 6 sessions. Each treatment session will last for a total of 45 minutes. A standardized physical therapy program will be used and will include soft tissue mobilization to the shoulder and biceps tendon and a standardized exercise program. Neither dry needling nor heavy slow load exercise will be integrated into the "control" plan of care. Participants will be instructed to do all activities that do not increase symptoms and avoid activities which aggravate symptoms as advice to maintain usual activity has been found to assist in recovery from shoulder pain. Both groups will be treated with a stretching and strengthening program. The rotator cuff and scapular stabilization strengthening and flexibility program

Individuals will complete the first 3 weeks of the study (either DN +HSLE or control) and will be asked to complete outcome measures (ASES, NPRS, DASH, SPADI, Medication usage, PSFS, GROC, PASS) at 3, 12 weeks, and 6 months, following the initiation of therapy for follow-up measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years old
* Primary diagnosis of bicipital tendinopathy
* Primary complaint of anterior shoulder pain in the area of the LHBT
* Clinical exam findings (must have positive findings for at least 1/2 of the following: Speed's Test, Yergason's test for biceps tendon pain.
* Pain with palpation in area of the biceps tendon
* Patient identification of pain in the area of the proximal biceps tendon
* NPRS of at least 3/10 at worst in the past week

Exclusion Criteria:

* History of biceps tendon injection in the past 3 months
* History of rotator cuff surgery
* History of biceps tenodesis or tenotomy
* History of bleeding disorder or anti-coagulation therapy
* Diagnosis of adhesive capsulitis (as defined by 50% loss of range of motion in 2 out of 3 of the following motions: Shoulder flexion, abduction and external rotation)
* Known underlying non-modifiable medical condition (e.g. tumor, fracture, metabolic disease)
* Two or more positive neurological signs consistent with nerve root compression
* Known allergy to metal
* Participant reported aversion to needles

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons Scale (ASES) at Baseline | Baseline
  shoulder pain and disability; The ASES is a 100-point shoulder-specific self-report questionnaire consisting of 2 subscales including pain and disability. Lower scores are indicative of higher levels of disability.
American Shoulder and Elbow Surgeons Scale (ASES) at 3 Weeks | 3 weeks
  shoulder pain and disability; The ASES is a 100-point shoulder-specific self-report questionnaire consisting of 2 subscales including pain and disability. Lower scores are indicative of higher levels of disability.
American Shoulder and Elbow Surgeons Scale (ASES) at 12 Weeks | 12 weeks
  shoulder pain and disability; The ASES is a 100-point shoulder-specific self-report questionnaire consisting of 2 subscales including pain and disability. Lower scores are indicative of higher levels of disability.
American Shoulder and Elbow Surgeons Scale (ASES) at 6 Months | 6 months
  shoulder pain and disability; The ASES is a 100-point shoulder-specific self-report questionnaire consisting of 2 subscales including pain and disability. Lower scores are indicative of higher levels of disability.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) at Baseline | Baseline
  Pain: An 11-point NPRS will be used to measure pain intensity. Numeric pain scales have been shown to be reliable and valid.61-65 Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. The average of the three ratings or any single rating may be used to represent the patient's level of pain.
Numeric Pain Rating Scale (NPRS) at 3 Weeks | 3 weeks
  Pain; An 11-point NPRS will be used to measure pain intensity. Numeric pain scales have been shown to be reliable and valid.61-65 Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. The average of the three ratings or any single rating may be used to represent the patient's level of pain.
Numeric Pain Rating Scale (NPRS) at 12 Weeks | 12 weeks
  Pain; An 11-point NPRS will be used to measure pain intensity. Numeric pain scales have been shown to be reliable and valid.61-65 Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. The average of the three ratings or any single rating may be used to represent the patient's level of pain.
Numeric Pain Rating Scale (NPRS) at 6 Months | 6 months
  Pain; An 11-point NPRS will be used to measure pain intensity. Numeric pain scales have been shown to be reliable and valid.61-65 Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. The average of the three ratings or any single rating may be used to represent the patient's level of pain.
DASH score at Baseline | Baseline
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH); The DASH is a 30 item, self-administered questionnaire that addresses symptoms and physical function in individuals with disorders of the upper limb.51 The DASH is scored from 0-100% (0% = no disability).
DASH score at 3 Weeks | 3 weeks
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH);The DASH is a 30 item, self-administered questionnaire that addresses symptoms and physical function in individuals with disorders of the upper limb.51 The DASH is scored from 0-100% (0% = no disability).
DASH score at 12 Weeks | 12 weeks
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH);The DASH is a 30 item, self-administered questionnaire that addresses symptoms and physical function in individuals with disorders of the upper limb.51 The DASH is scored from 0-100% (0% = no disability).
DASH score at 6 Months | 6 months
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH);The DASH is a 30 item, self-administered questionnaire that addresses symptoms and physical function in individuals with disorders of the upper limb.51 The DASH is scored from 0-100% (0% = no disability).
Patient specific functional scale (PSFS) at Baseline | Baseline
  Patient assessment of function; The PSFS is a patient self-reported measurement tool used to assess functional change. Patients identify up to 5 activities at Baseline that they find difficult or impossible to perform due to their problem, and then rate the difficulty level of each activity from 0 (unable to perform) to 10 (able to perform activity at same level as before injury/problem). The sum of the 5 scores will be reported and assessed for change at subsequent timepoints
Patient specific functional scale (PSFS) at 3 Weeks | 3 weeks
  Patient assessment of function; The PSFS is a patient self-reported measurement tool used to assess functional change. Patients identify up to 5 activities at Baseline that they find difficult or impossible to perform due to their problem, and then rate the difficulty level of each activity from 0 (unable to perform) to 10 (able to perform activity at same level as before injury/problem). The sum of the 5 scores will be reported and assessed for change at subsequent timepoints
Patient specific functional scale (PSFS) at 12 Weeks | 12 weeks
  Patient assessment of function; The PSFS is a patient self-reported measurement tool used to assess functional change. Patients identify up to 5 activities at Baseline that they find difficult or impossible to perform due to their problem, and then rate the difficulty level of each activity from 0 (unable to perform) to 10 (able to perform activity at same level as before injury/problem). The sum of the 5 scores will be reported and assessed for change at subsequent timepoints
Patient specific functional scale (PSFS) at 6 Months | 6 months
  Patient assessment of function; The PSFS is a patient self-reported measurement tool used to assess functional change. Patients identify up to 5 activities at Baseline that they find difficult or impossible to perform due to their problem, and then rate the difficulty level of each activity from 0 (unable to perform) to 10 (able to perform activity at same level as before injury/problem). The sum of the 5 scores will be reported and assessed for change at subsequent timepoints
Global Rating of Change (GROC) at 3 Weeks | 3 weeks
  Patient perceived level of change; The fifteen-point global rating scale described by Jaeschke et al. will be used.53 The scale ranges from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). Descriptors of worsening or improving are assigned values from -1 to -6 and +1 to +6 respectively.
Global Rating of Change (GROC) at 12 Weeks | 12 weeks
  Patient perceived level of change; The fifteen-point global rating scale described by Jaeschke et al. will be used.53 The scale ranges from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). Descriptors of worsening or improving are assigned values from -1 to -6 and +1 to +6 respectively.
Global Rating of Change (GROC) at 6 Months | 6 months
  Patient perceived level of change; The fifteen-point global rating scale described by Jaeschke et al. will be used.53 The scale ranges from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). Descriptors of worsening or improving are assigned values from -1 to -6 and +1 to +6 respectively.
Medication Usage at Baseline | baseline
  Use of medication; medication name, dose and frequency per day/week will be tracked
Medication Usage at 3 Weeks | 3 weeks
  Use of medication; medication name, dose and frequency per day/week will be tracked
Medication Usage at 12 Weeks | 12 weeks
  Use of medication; medication name, dose and frequency per day/week will be tracked
Medication Usage at 6 Months | 6 months
  Use of medication; medication name, dose and frequency per day/week will be tracked
Should Pain and Disability Index | Baseline
  participant report of shoulder related pain and disability (how shoulder pain limits function)
Should Pain and Disability Index | 3 weeks
  participant report of shoulder related pain and disability (how shoulder pain limits function)
Should Pain and Disability Index | 12 weeks
  participant report of shoulder related pain and disability (how shoulder pain limits function)
Should Pain and Disability Index | 6 months
  participant report of shoulder related pain and disability (how shoulder pain limits function)

CONTACTS AND LOCATIONS:
Overall Officials: Amy W McDevitt, DPT, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Education 1 Anschutz Medical Campus, Aurora, Colorado
  - Boulder Center for Sports Medicine and Performance, Boulder, Colorado

IPD SHARING:
Plan to Share IPD: No
There is not a plan at this time